CLINICAL TRIAL: NCT03133754
Title: Open-lung Ventilatory Approach With Positive End-expiratory Pressure Titrated to Lowest Driving Pressure in Cardiac Surgery Patients
Brief Title: OLA to Lowest DP in Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Principal Investigator, Carlos Ferrando, Principal investigador, Fundación para la Investigación del Hospital Clínico de Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DP-PEEP
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Lung Collapse
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DP-PEEP (Experimental): recruitment maneuver + individualized PEEP
  Interventions: Procedure: DP-PEEP
- RM-5 (Active Comparator): recruitment maneuver + fixed standard PEEP
  Interventions: Procedure: RM-5

INTERVENTIONS:
Procedure: DP-PEEP — PEEP titration trial for the lowest DP after the alveolar recruitment maneuver
  Arms: DP-PEEP
Procedure: RM-5 — Fixed standard PEEP after the alveolar recruitment maneuver
  Arms: RM-5

SUMMARY:
This study aims to compared the effects in driving pressure of an open-lung strategy with a positive end-expiratory pressure (PEEP) titrated to best driving pressure (DP) after a RM versus the recommended protective PEEP of 5 cmH2O without a recruitment manuever in non-obese patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Non-obese patients scheduled for cardiac surgery (CABG and valve replacement)

Exclusion Criteria:

* i) age <18yr or >80yr, ii) pregnancy or breast-feeding status, and iii) patients with previous known respiratory disease, iv) Body mass index >35 kg/m2, v) emergency surgery and vi) hemodynamic instability at entry (need of vasopressors or ionotropes at entry or a ventricular assist device.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
driving pressure | intraoperative
  The driving pressure is a physiological ventilatory parameter measured as platteau pressure minus PEEP. This parameter may be associated with postoperative pulmonary complications

SECONDARY OUTCOMES:
Postoperative pulmonary complications | 72 first postoperative hours
  The most frequent postoperative pulmonary complications will be recorded (acute respiratory failure, pneumonia, atelectasis, need of ventilatory support, acute respiratory distress syndrome)

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos Ferrando, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Costa Leme A, Hajjar LA, Volpe MS, Fukushima JT, De Santis Santiago RR, Osawa EA, Pinheiro de Almeida J, Gerent AM, Franco RA, Zanetti Feltrim MI, Nozawa E, de Moraes Coimbra VR, de Moraes Ianotti R, Hashizume CS, Kalil Filho R, Auler JO Jr, Jatene FB, Gomes Galas FR, Amato MB. Effect of Intensive vs Moderate Alveolar Recruitment Strategies Added to Lung-Protective Ventilation on Postoperative Pulmonary Complications: A Randomized Clinical Trial. JAMA. 2017 Apr 11;317(14):1422-1432. doi: 10.1001/jama.2017.2297. PMID 28322416
- [Background] Serpa Neto A, Hemmes SN, Barbas CS, Beiderlinden M, Biehl M, Binnekade JM, Canet J, Fernandez-Bustamante A, Futier E, Gajic O, Hedenstierna G, Hollmann MW, Jaber S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Putensen C, Ranieri M, Scavonetto F, Schilling T, Schmid W, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Gama de Abreu M, Pelosi P, Schultz MJ; PROVE Network Investigators. Protective versus Conventional Ventilation for Surgery: A Systematic Review and Individual Patient Data Meta-analysis. Anesthesiology. 2015 Jul;123(1):66-78. doi: 10.1097/ALN.0000000000000706. PMID 25978326
- [Background] Ferrando C, Soro M, Canet J, Unzueta MC, Suarez F, Librero J, Peiro S, Llombart A, Delgado C, Leon I, Rovira L, Ramasco F, Granell M, Aldecoa C, Diaz O, Balust J, Garutti I, de la Matta M, Pensado A, Gonzalez R, Duran ME, Gallego L, Del Valle SG, Redondo FJ, Diaz P, Pestana D, Rodriguez A, Aguirre J, Garcia JM, Garcia J, Espinosa E, Charco P, Navarro J, Rodriguez C, Tusman G, Belda FJ; iPROVE investigators (Appendices 1 and 2). Rationale and study design for an individualized perioperative open lung ventilatory strategy (iPROVE): study protocol for a randomized controlled trial. Trials. 2015 Apr 27;16:193. doi: 10.1186/s13063-015-0694-1. PMID 25927183
- [Background] Borges DL, Nina VJ, Costa Mde A, Baldez TE, Santos NP, Lima IM, Figueredo ED, Lula JL. Effects of different PEEP levels on respiratory mechanics and oxygenation after coronary artery bypass grafting. Rev Bras Cir Cardiovasc. 2013 Jul-Sep;28(3):380-5. doi: 10.5935/1678-9741.20130058. PMID 24343688
- [Background] Reis Miranda D, Gommers D, Struijs A, Dekker R, Mekel J, Feelders R, Lachmann B, Bogers AJ. Ventilation according to the open lung concept attenuates pulmonary inflammatory response in cardiac surgery. Eur J Cardiothorac Surg. 2005 Dec;28(6):889-95. doi: 10.1016/j.ejcts.2005.10.007. Epub 2005 Nov 3. PMID 16271479